CLINICAL TRIAL: NCT02121379
Title: Randomized Clinical Trial of 8 Weeks Pulmonary Rehabilitation in Advanced Stage Lung Cancer Patients With COPD During Cytotoxic Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young Sik Park, Assitant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1401-116-549
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: COPD; Lung Cancer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

ARMS (2):
- control (No Intervention): stretching exercise
- pulmonary rehablitation (Experimental): warming up exercise strengthening exercise aerobic exercise cool down
  Interventions: Behavioral: pulmonary rehabilitation

INTERVENTIONS:
Behavioral: pulmonary rehabilitation
  Arms: pulmonary rehablitation

SUMMARY:
Pulmonary rehabilitation might be benificial in advanced lung cancer patients with COPD who undergo cytotoxic chemotherapy.

We will compare two groups, 8 week pulmonary rehabilitation group and usual care group.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven lung cancer
* chronic obstructive pulmonary disease
* age > 20
* ECOG 0-1
* cytotoxic chemotherapy

Exclusion Criteria:

* other history of cancer within 5 years
* other major disease associated with heart, lung, neurology, mental and metabolic disorders
* osteolytic bone metastatis to weight bearing site
* uncontrolled infection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
difference of VO2 max | 8 weeks
  difference maximal oxygen consumption during exercise cardiopulmonary test between before and after intervention/control

SECONDARY OUTCOMES:
difference of Saint George's Respiratory Questionannaire (SGRQ) score | 8 weeks
  the difference of SGRQ score
difference of pulmonary function test | 8 weeks
  the difference of FVC and FEV1
difference of 6 min walk test | 8 weeks
  the difference of 6 minute walk test
difference of depression test | 8 weeks
  using Hospital Anxiety and Depression scale (HADS), measure the difference HADS between before and after intervention/control

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea